CLINICAL TRIAL: NCT05729750
Title: Efficacy of Music Listening to Shortening Time for Biophysical Profile
Acronym: RRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 004/2565
Record Dates: First submitted 2023-01-04; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-12

CONDITIONS: Fetal Status, Nonreassuring
Keywords: Fetal biophysical profile; Music; Duration
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Intervention Model Description: the participants were purpostive sampling, and devided into two groups. The study group listening to music before and suring the assessment while the control gruop will not listening to music.
Who Masked: Investigator
Masking Description: All participants whatever study or control gruops will get the headphone which may turn on the music in study gruop only that mean investigator will not known who are in listening to music.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lable litter A (Study group) (Experimental): The sealed opaque brown envelope contains a case record form and the letter A paper for listening to the music before and during the BPP assessment (study group), which cannot be visible from the outside.
  Interventions: Diagnostic Test: Trans abdominal ultrasound for assess biophysical profile
- Lable litter B (control group) (Placebo Comparator): The sealed opaque brown envelope contains a case record form and the letter B for not listening to the music before and during the BPP assessment (control group), which cannot be visible from the outside.
  Interventions: Diagnostic Test: Trans abdominal ultrasound for assess biophysical profile

INTERVENTIONS:
Diagnostic Test: Trans abdominal ultrasound for assess biophysical profile — The biophysical profile (BPP) was developed as a method of integrating real-time observation of the fetus in an intrauterine environment. Manning et al introduced the BPP test in 1980, and since then it has been widely used as a comprehensive assessment tool for both acute and chronic fetal health and fetal congenital malformations in the antepartum period which is a method that uses an overview of 5 key indicators, namely fetal tone, fetal breathing, fetal movement, deep ventricular pocket and NST, thus making it more accurate than either viewing.

SUMMARY:
The goal of this clinical trial is to compare the timeing which assume for assesment of BPP in low risk pregnancy. The main question is the music can be shoetening the timing for BPP? Participants will in study froup will listening the music via headphone before and during the assessment and compre to control gruop which not listening to music during asseeement.

DETAILED DESCRIPTION:
A single-blind randomized controlled trial conducted from February 2021 to December 2022. The study population consisted of 60 pregnant women with between 18 and 35 years old with gestational age of 32 weeks. An abdominal ultrasound was performed while listening to one song while wearing headphones in the experimental group preceding the biophysical profile assessment. As part of the control group, the same equipment was used and the same assessment protocol was followed, but music was not played during the test.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy (Singleton)
* Gestational age from 32 weeks onward
* Pregnant women do not have underlying diseases such as pre-gestational diabetes. high blood pressure
* No abnormalities in the fetus were found, such as fetal deformities.

Exclusion Criteria:

* Pregnant women receiving certain drugs or substances that affect the interpretation of the Biophysical Profile (BPP), e.g., sleeping pills, cigarettes.
* Pregnant women have hearing problems. or hearing impaired
* Pregnant women who are unable to wear headphones, e.g., otitis externa - Pregnant women with body mass index greater than 30 kg/m2 prior to pregnancy
* Uterine contractions were observed during the examination

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnants woman
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Total time used for the biophysical profile | Through study complete, an average 30 minutes
  To compare the total time of biophysical profile assessment among pregnant women listening to music or not listening to music

SECONDARY OUTCOMES:
Satisfaction of music | After study complete, an average 30 minutes
  To measure music listening satisfaction in experimental groups on a scale of 1 (unsatisfied) to 5 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Bhanubhan Meepon, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data was save inform of microsoft excel spreadsheet and SPSS file.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From march 2023
URL: https://1drv.ms/x/s!Aiv4SoaNlXd8k2mwfx0qeh0g1DLC